CLINICAL TRIAL: NCT01363557
Title: Randomized to Assess the Efficacy of Whole Brain Radiation Therapy (WBRT) With Concomitant Gefitinib Followed by Maintenance Gefitinib, and Gefitinib Alone, in Lung Cancer Patients With Brain Metastasis
Brief Title: Assess the Efficacy of Whole Brain Radiation Therapy in Lung Cancer Patients With Brain Metastasis
Acronym: ARPEGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of Sponsor
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100601; 2010-A01332-37 (Other: IDRCB)
Record Dates: First submitted 2011-05-25; First posted 2011-06-01 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: EGFR-mutated Lung Adenocarcinoma; Brain Metastasis
Keywords: Randomized; Brain Radiation Therapy; Lung Cancer; Brain Metastasis; Gefitinib
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A : Gefitinib + WBRT (Experimental): Arm A : WBRT and Concurrent Gefitinib followed by Gefitinib Maintenance
  Interventions: Other: whole brain radiotherapy
- Arm B : Gefitinib (Experimental): Arm B : Gefitinib alone
  Interventions: Drug: Gefitinib (IRESSA)

INTERVENTIONS:
Other: whole brain radiotherapy — External beam RT using a total dose of 30 Gy with ten daily fractions of 3.0 Gy given 5 days per week over 2 weeks + Gefitinib 250 mg/day
  Arms: Arm A : Gefitinib + WBRT
Drug: Gefitinib (IRESSA) — 250 mg/day
  Arms: Arm B : Gefitinib

SUMMARY:
Multicentre randomised (1:1) trial assessing the efficacy of whole brain radiotherapy in addition to Gefitinib for the management of brain metastasis in lung cancer patients with a mutated EGFR.

DETAILED DESCRIPTION:
Lung cancer patients with newly diagnosed CNS metastasis with- at least one brain lesion measuring > 1 cm in longest dimension - not eligible for surgery or stereotactic radio-surgeryOpen-label, multicentre, national, randomised (1:1) phase II trialArm A: WBRT and Concurrent Gefitinib followed by Gefitinib Maintenance Arm B: Gefitinib

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed a written informed consent form prior to any study specific screening procedures
* 18 years or older
* KPS ≥ 50%
* Histologically confirmed adenocarcinoma of the lung
* Activating mutation of EGFR
* Newly diagnosed CNS metastasis or in progression with at least one measurable lesion in the brain (defined as any lesion > 1 cm on T1-weighted contrast enhanced MRI)
* Patients could enter the study regardless of previous treatment (included chemotherapy) for metastatic extracranial disease, except TKI.
* No steroids or stable or decreasing dose of steroids for at least 5 days before the MRI evaluation.
* Adequate hematologic, liver and renal functions: neutrophil count ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; Hb ≥ 9 g/Dl; Total bilirubin < 1.5 x ULN; AST or ALT < 2.5 x ULN (< 5 x ULN in patients with liver metastases); Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* Prior treatment of brain metastases with WBRT or TKI
* Patient eligible for radiosurgery or surgical resection
* Contre indication at the radiotherapy
* Leptomeningeal disease
* Previous history of cancer (other than curatively treated basal and squamous cell carcinoma of the skin and/or in-situ carcinoma of the cervix) within the the 5 years before study entry
* Prior treatment with Gefitinib or other TKI
* Pregnant or breast feeding women
* Women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To assess the objective response rate of brain metastases in each arm | at 6 weeks

SECONDARY OUTCOMES:
Number of Participants with neurological Adverse Events | at 6 weeks, 3 months, 4.5 months and 6 months
Progression-free survival (PFS) | at 6 months
Overall survival | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CARPENTIER, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Neurologie - Hôpital Avicenne, Bobigny, France